CLINICAL TRIAL: NCT05709093
Title: A Randomized, Controlled, Open-label, Multicenter Phase 3 Clinical Study to Evaluate Lemzoparlimab for Injection in Combination With Azacitidine (AZA) Versus AZA Monotherapy in Treatment-naïve Patients With Higher-risk Myelodysplastic Syndrome (MDS)
Brief Title: A Phase 3 Clinical Study to Evaluate Lemzoparlimab for Injection in Combination With Azacitidine (AZA) Versus AZA Monotherapy in Treatment-naïve Patients With Higher-risk Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company Development strategy adjustment]
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ011133MDS301
Record Dates: First submitted 2023-01-10; First posted 2023-02-01 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Myelodysplastic Syndromes(MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lemzoparlimab in combination with AZA (Experimental)
  Interventions: Drug: Lemzoparlimab+Azacitidine (AZA)
- AZA monotherapy (Active Comparator)
  Interventions: Drug: Azacitidine (AZA)

INTERVENTIONS:
Drug: Lemzoparlimab+Azacitidine (AZA) — 1. Lemzoparlimab is administered by intravenous (IV) infusion once a week at a dose of 30 mg/kg in 28-day treatment cycles
  2. Azacitidine (AZA): AZA is administered by subcutaneous injection once a day at a dose of 75 mg/m2 on D1 to D7 of each treatment cycle in 28-day treatment cycles.
  Arms: Lemzoparlimab in combination with AZA
Drug: Azacitidine (AZA) — AZA is administered by subcutaneous injection once a day at a dose of 75 mg/m2 on D1 to D7 of each treatment cycle in 28-day treatment cycles.
  Arms: AZA monotherapy

SUMMARY:
This phase3 study is a randomized, controlled, open-label, multicenter study to evaluate the efficacy and safety of Lemzoparlimab for injection in combination with AZA versus AZA monotherapy as first-line therapy in treatment-naïve subjects with intermediate- and high-risk MDS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 18 years of age at the time of signing the ICF.
* Subjects with intermediate- and high-risk MDS who are confirmed by bone marrow aspiration or pathological biopsy according to the diagnostic criteria of World Health Organization (WHO) 2016 or who are eligible for blasts in bone marrow and peripheral blood < 20% and have a score > 3.5 according to the revised International Prognostic Scoring System (IPSS-R).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2.
* Subjects without any prior anti-tumor therapy for MDS, including demethylated drugs (eg, AZA, decitabine), chemotherapy, targeted therapy, or HSCT. The blood transfusion or use of hematopoietic growth factors and supplementation of hematopoietic raw materials such as folic acid, vitamin B12 are permitted. For patients who ever took lenalidomide, thalidomide, antithymocyte globulin (ATG), or ciclosporin before study entry, there should be a washout period of at least 28 days prior to the first dose.
* Subjects who are eligible for HSCT and have no pre-scheduled HSCT at screening, or subjects who are ineligible for HSCT and have no scheduled HSCT at screening
* Expected survival ≥ 12 weeks
* Subjects with adequate organ function and laboratory tests meet the following requirements
* Female subjects of childbearing potential or male subjects whose partner is a woman of childbearing potential are required to use effective contraception throughout the treatment period and until 6 months after the treatment period.
* Subjects must be willing to provide available diagnostic evidence or undergo bone marrow aspiration and biopsy before study treatment, and must be willing to undergo bone marrow aspiration and biopsy after receiving study treatment.
* Subjects must give informed consent before starting the study and sign written ICF voluntarily by themselves (or their legal representatives). Subjects or their legal representatives should be able to communicate well with investigators and agree to adhere with the study protocol and complete the study

Exclusion Criteria:

* Patients who have transformed from MDS to AML, or have been diagnosed with treatment-related MDS (t-MDS), or patients with myeloproliferative neoplasia (MPN) or myelodysplastic syndrome/myeloproliferative disorder (MDS/MPN) that meet WHO 2016 criteria
* Previously received any anti-CD47 antibody or SIRPα antibody or the drugs targeting the same target
* Subjects have received or plan to receive the allogeneic stem cell transplantation or organ transplantation during the study
* History of chronic hemolytic anemia due to other diseases or clinically significant positive hemolysis-related test at screening (except positive hemolysis test due to MDS)
* Concurrent participation in another interventional clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Subjects plan to receive other anti-tumor therapies, including but not limited to chemotherapy, biotherapy and immunotherapy, while participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival Overall Survival(OS) | From date of randomization until the date of first documented progression or date from any cause,whichever came first, assessed up to 50 months.

CONTACTS AND LOCATIONS:
Locations (44):
- China (44):
  - The First Affiliated Hospital Of Bengbu Medical College, Bengbu, Anhui
  - The First Affilated Hospital Of USTC Anhui Provincial Hospital, Hefei, Anhui
  - THE First Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - Beijing Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Gaobo Boren Hospital Co., Ltd, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of PLA Army Military Medical University, Chongqing, Chong Qing
  - The Second Affiliated Hospital of Army Medical University, Chongqing, Chong Qing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chong Qing
  - The Affiliated Zhongshan Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Southern Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Harbin First Hospital, Harbin, Heilongjiang
  - First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Medical College of HUST, Wuhan, Hubei
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Changsha Third Hospital, Changsha, Hunan
  - The Affiliated Hosptial Of XuZhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shaanxi Provincial People's Hospital, Xi'an, Shaan XI
  - The Second Affiliated Hospital of Xi'an Jiaotong University Medical College, Xi'an, Shaanxi
  - Cheeloo College of Medicine, Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Tai’an, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Renji Hospital Affiliated to Medical College of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang
  - The First Affiliated Hospital Of WenZhou Medical College, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided